CLINICAL TRIAL: NCT01539811
Title: Surgical Management of Diabetic Foot Infections - The Role of Post-Operative Antibiotics
Brief Title: Diabetic Foot Infection Antibiotic Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator decided to terminate the study.
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00015080
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Foot Infections
Keywords: Foot Infections; Diabetes; Antibiotic
MeSH Terms: conditions — Diabetes Mellitus | interventions — Amputation, Surgical; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short course antibiotics (Active Comparator): Surgical intervention followed by short course of antibiotics (<2 weeks)
  Interventions: Procedure: Surgical incision and drainage of diabetic foot infection; Drug: Short course antibiotics
- Long course antibiotics (Active Comparator): Surgical intervention followed by a long course of antibiotics (>2 weeks)
  Interventions: Procedure: Surgical incision and drainage of diabetic foot infection; Drug: Long course antibiotics

INTERVENTIONS:
Procedure: Surgical incision and drainage of diabetic foot infection — Incision and drainage of diabetic foot infection with or without amputation of toes or the forefoot, depending on the condition of the foot
  Other Names: Surgical debridement; Bone resection; Amputation
Drug: Short course antibiotics — Short course (<2 weeks) of antibiotics will be prescribed
  Other Names: IV antibiotics; oral antibiotics
  Arms: Short course antibiotics
Drug: Long course antibiotics — Long course (>2 weeks) of antibiotics will be prescribed
  Other Names: IV antibiotics; oral antibiotics
  Arms: Long course antibiotics

SUMMARY:
This is a pilot study to explore the effects of long-course versus short course antibiotics on wound healing in surgically managed diabetic foot infections. Hypothesis: Diabetic Foot Infections (DFIs) are best managed with an early aggressive surgical approach and short term antibiotic use. Post-operative prolonged antibiotic use increases costs and resource utilization without improving outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to optimize the management of diabetic foot infections. In this cost conscious health care environment, we believe that equal outcomes can be obtained through more cost effective and efficient means. In order to conduct more definitive studies of the role of antibiotic therapy regimens in diabetic foot infections, we first must collect pilot data to determine both the feasibility and most appropriate methods (sample size, etc.) for designing these larger trials.

Currently, the best way to manage these infections remains elusive; many studies suggest medical management is sufficient with surgical management reserved for failure of medical management or aggressive foot infections; however, this approach leads to recurrence and delays definitive treatment at a significant increase in costs. Several meta-analysis studies have tried to find the best antibiotic regimen; however, due to the vast discrepancies in study design and endpoints no conclusive evidence exists for which is the best antibiotic regimen in patients treated medically, let alone patients with more complicated disease whom require surgical management.

The Infectious Diseases Society of America (IDSA) guidelines have provided recommendations; however, the optimal length is not standardized and to date no studies have looked at the best regimen for post-operative management of surgically treated diabetic foot infections and whether antibiotics help in the healing process. The IDSA guideline suggest that antibiotics are necessary for virtually all infected wounds, but specific guidance for surgically treated wounds is lacking.

This is a randomized, single-blinded study (Infectious disease physicians whom will determine long-term treatment will be blinded). Randomization will occur by blocked random allocation scheme using randomization software and a block size of 10. The study coordinator will keep the randomization schedule/log and inform the surgeon which therapy the patient will receive

* Treatment group #1: Surgical intervention, short term course of antibiotics (< 2 week post-op)
* Treatment group #2: Surgical intervention, long term course of antibiotics (> 2 week post-op)

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment for moderate (Grade 3-IDSA guidelines) infection of one or more toes from diabetes mellitus

Exclusion Criteria:

* IDSA Grade 1,2, or 4 infections
* Non-diabetic foot ulcers
* Non-infected foot ulcers
* Sepsis
* Currently taking antibiotics for reasons not related to foot infection
* Infections requiring a transmetatarsal amputation
* Ischemic ulcers
* Gangrene
* Revascularization within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Cull, M.D., Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Hospital System University Medical Center, Greenville, South Carolina, United States

REFERENCES:
- [Background] Armstrong DG, Lipsky BA. Diabetic foot infections: stepwise medical and surgical management. Int Wound J. 2004 Jun;1(2):123-32. doi: 10.1111/j.1742-4801.2004.00035.x. PMID 16722884
- [Background] Joseph WS, Lipsky BA. Medical therapy of diabetic foot infections. J Vasc Surg. 2010 Sep;52(3 Suppl):67S-71S. doi: 10.1016/j.jvs.2010.06.010. PMID 20804935
- [Background] Fisher TK, Scimeca CL, Bharara M, Mills JL Sr, Armstrong DG. A step-wise approach for surgical management of diabetic foot infections. J Vasc Surg. 2010 Sep;52(3 Suppl):72S-75S. doi: 10.1016/j.jvs.2010.06.011. PMID 20804936
- [Background] Lipsky BA, Holroyd KJ, Zasloff M. Topical versus systemic antimicrobial therapy for treating mildly infected diabetic foot ulcers: a randomized, controlled, double-blinded, multicenter trial of pexiganan cream. Clin Infect Dis. 2008 Dec 15;47(12):1537-45. doi: 10.1086/593185. PMID 18990064
- [Background] Margolis DJ, Gelfand JM, Hoffstad O, Berlin JA. Surrogate end points for the treatment of diabetic neuropathic foot ulcers. Diabetes Care. 2003 Jun;26(6):1696-700. doi: 10.2337/diacare.26.6.1696. PMID 12766096
- [Background] Stoner MC, Defreitas DJ, Manwaring MM, Carter JJ, Parker FM, Powell CS. Cost per day of patency: understanding the impact of patency and reintervention in a sustainable model of healthcare. J Vasc Surg. 2008 Dec;48(6):1489-96. doi: 10.1016/j.jvs.2008.07.003. Epub 2008 Oct 1. PMID 18829227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Course Antibiotics | Long Course Antibiotics
Started | 0 (Antibiotics never given. Study closed prior to initiating treatment.) | 0 (Antibiotics never given. Study closed prior to initiating treatment.)
Completed | 0 (Antibiotics never given. Study closed prior to initiating treatment.) | 0 (Antibiotics never given. Study closed prior to initiating treatment.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Both enrolled patients were deemed ineligible soon after enrollment and therefore participants analyzed were zero
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Course Antibiotics | Long Course Antibiotics | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing
Description: Wound healing at 3 months (75% epithelialization) from the time of the final definitive operation.
Time Frame: 3 months
Population: study closed with only 2 patient enrolled, who were both deemed ineligible prior to the outcome measure window. No patients reached the 3 month time period for the outcome measure.
Arm/Group | Short Course Antibiotics | Long Course Antibiotics
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The 2 enrolled patients were deemed ineligible shortly after enrollment, prior to implementation of randomized treatments (<2 weeks), prior to collection of any Adverse events.
Arm/Group | Short Course Antibiotics | Long Course Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No